CLINICAL TRIAL: NCT07084155
Title: Adaptive Cell Phone Support to Promote Medication Adherence Among Adolescents and Young Adults With Chronic Health Conditions
Brief Title: Final Prototype Refinement of Adaptive Cell Phone Support
Acronym: ACPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Caitlin Sayegh, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-23-00149_Phase II
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Medication Adherence
Keywords: adolescents; mobile health; adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adaptive Cell Phone Support (Experimental): Computer-delivered cell phone support (reminders, problem-solving, referrals to resources) and responsive human coaching (phone calls, test messages, in-app messaging) to improve medication adherence.
  Interventions: Behavioral: Adaptive Cell Phone Support

INTERVENTIONS:
Behavioral: Adaptive Cell Phone Support — Mobile health adherence promotion based on the supportive accountability model

SUMMARY:
The goal of this feasibility pilot trial is to finalize the design of a mobile health intervention for promoting medication adherence in a population of adolescents and young adults with chronic health conditions. The main question[s] it aims to answer are:

1. Is the final version of the intervention sufficiently feasible, usable, and acceptable for evaluation in a randomized clinical trial?
2. Do participants show improvements in medication adherence during their field testing of the intervention?

DETAILED DESCRIPTION:
Adolescents with chronic health conditions will be asked to try the intervention for three weeks and give feedback to refine the structure and content in preparation for a future randomized trial of the finalized version of the intervention. Plan to enroll 35 participants in this single arm feasbility/usability trial.

ELIGIBILITY:
Inclusion Criteria:

* Children's Hospital Los Angeles patient
* between 15-20 years old
* taking at least one oral medication per day for a chronic health condition
* English speaking
* demonstrating sufficient cognitive capacity to engage in the assent/consent process and study procedures

There is no exclusion criteria.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Total scores on the theoretical framework of acceptability questionnaire | Baseline to 3 weeks
  Higher scores indicate a greater "extent to which people delivering or receiving a healthcare intervention consider it to be appropriate, based on anticipated or experienced cognitive and emotional responses to the intervention"; the minimum value of this questionnaire is 7 and the maximum value is 35.
Mean scores on the Mobile Health App Usability Questionnaire | Baseline to 3 weeks
  Higher scores indicate greater ease with which users can use technology to achieve a particular goal; the minimum value of this questionnaire is 1 and the maximum value is 7.
Total scores on the Visual Analogue Scale | Baseline to 3 weeks
  Percentage of doses taken our of 100%; higher numbers indicate greater medication adherence. This scale presents participants with a line, marked 0 on the left and 100 on the right, and participants can drag a marker to the place on the line that best visually indicated their adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Sayegh, PhD, Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: Yes
The data will include electronically-administered survey items assessing demographic characteristics, intervention usability, intervention acceptability, medication adherence, motivation for adherence, transition readiness skills, and allocation of treatment responsibility as well as medication regimen complexity data and pharmacy possession refill rates abstracted from the electronic medical chart, and behavioral engagement data collected via the Computerized Intervention Authoring Software.
Time Frame: Final submission and release of the study data will occur no later than the time of an associated publication or the end of the performance period, whichever comes first. Study data deposited in DASH will be available to the research community in perpetuity.
Access Criteria: https://dash.nichd.nih.gov/resource/DASHUserAgreement
URL: https://dash.nichd.nih.gov/